CLINICAL TRIAL: NCT04827290
Title: Assessment of the Effect of Restriction on Alimentary AGE (Advanced Glycation Products) in Progression of Chronic Kidney Disease (CKD)
Brief Title: Assessment of the Effect of Restriction on Alimentary AGE in Progression of Chronic Kidney Disease
Acronym: CKD AGE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Saint Joseph Saint Luc de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CKD AGE
Record Dates: First submitted 2021-03-30; First posted 2021-04-01 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Kidney Failure, Chronic; Chronic Kidney Disease stage3; Chronic Kidney Disease Stage 3B; Chronic Kidney Disease Stage 3A (Disorder); Chronic Kidney Disease, Stage 3 (Moderate); Diet Habit
Keywords: kidney failure; advanced glycation products; chronic kidney disease
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic; Lymphoma, Follicular; Feeding Behavior; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal-protein and low-AGE through raw or rare proteins diet (Experimental): Normal-protein (0,8g/kg/day) and low-AGE through raw or rare proteins diet during 24 months
  Interventions: Behavioral: Low-AGE diet
- Normal-protein and AGE-rich diet (Active Comparator): Normal-protein (0,8g/kg/day) and high-AGE through overcooked proteins diet during 24 months
  Interventions: Behavioral: High-AGE diet

INTERVENTIONS:
Behavioral: Low-AGE diet — Low-AGE diet during 24 months
  Arms: Normal-protein and low-AGE through raw or rare proteins diet
Behavioral: High-AGE diet — High-AGE diet during 24 months
  Arms: Normal-protein and AGE-rich diet

SUMMARY:
Normal-protein and low-AGE through raw or rare proteins diet versus normal-protein and high-AGE diet in stage IIIa-b renal failure patients

ELIGIBILITY:
Inclusion Criteria:

* Patients with a grade IIIA-B CKD (GFR with CKD-EPI ≥ 30 mL/min and < 60mL/min)
* Informed consent signed
* Aged 18 to 89 years

Exclusion Criteria:

* Protected adult
* Acute renal failure
* Patient already on a low-AGE diet (< 1kU AGE/day) following a dietetic consultation
* Current participation in another interventional research

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Glomerular Filtration Rate | At 24 months
  Glomerular Filtration Rate estimated by the CKD-EPI formula with a blood sample

SECONDARY OUTCOMES:
Proteinuria | At 24 months
  Proteinuria (g/24h) found in the 24-hour urine

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Saint Joseph Saint Luc, Lyon, France

IPD SHARING:
Plan to Share IPD: No